CLINICAL TRIAL: NCT05365763
Title: Developing an Experimental Framework to Evaluate Oncologist Emotion Regulation and Its Effect on Prognostic Disclosure During Telehealth Encounters
Brief Title: Developing an Experimental Framework to Evaluate Oncologist Emotion Regulation
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Garrett T. Wasp, Assistant Professor, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02000696
Record Dates: First submitted 2021-10-14; First posted 2022-05-09 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Communication
Keywords: serious illness conversation; serious illness communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical oncologists: 5 medical oncologists; trained in the serious illness conversation guide
  Interventions: Behavioral: Simulated telehealth serious illness conversation visit
- specialty palliative care: 6 specialty palliative care physicians; trained in serious illness conversation guide
  Interventions: Behavioral: Simulated telehealth serious illness conversation visit

INTERVENTIONS:
Behavioral: Simulated telehealth serious illness conversation visit — The study team will instruct the participant to relax, and record biometric data for a total 7 minutes (the beginning two minutes is to allow for physiologic adaptation).
  Simulated Encounter The study team will train experienced actors in the same case, a patient with a metastatic soft tissue sarcoma already on second-line chemotherapy. The physicians will receive a simulated medical file that contains a prognosis in a single format: a range-based, time prognosis (e.g. months to a year). The actor script and medical file will be developed by a multidisciplinary team (e.g. oncologist, palliative care, emotion scientist). The encounter will occur via tele-video platform (ZOOM®) and will be video-recorded. During the encounter participant physicians will wear three biometric sensors.

SUMMARY:
The research team recruited physicians (medical oncologists and specialty palliative care providers) trained in a communication tool called the serious illness conversation guide. Physicians conducted a simulated, telehealth serious illness conversation with an actor playing the role of a patient with advanced cancer. Physicians completed psychologic inventories before and after the encounter, documented the encounter using a template in the electronic medical record, and then participated in a structured interview afterwards discussing what they were feeling during the encounter and how it impacted the encounter. Physicians also wore three heart rate variability sensors during the simulated encounter.

DETAILED DESCRIPTION:
Aim 1: Assess the feasibility and acceptability of measuring physician emotion regulation (ER) abilities and strategies when disclosing prognosis in a simulated, outpatient telehealth encounter with a patient with advanced cancer.

This works seeks to address a technical gap in measurement relevant to the field of serious illness communication by assessing the feasibility and acceptability of collecting psychologic inventories and physiologic data in clinicians during a simulated patient encounter. The research team will purposely recruit physician of varied communication skill, assess communication behavior and triangulate different measures of emotion and ER (e.g. self-report, observation and biometric data sources). This exploratory aim will provide information regarding the feasibility of collecting data from physicians, variability in predictor (ER abilities) and outcome (prognostic disclosure and responding to patient emotion) measures, and preliminarily assess the construct validity of novel measures of physician ER. The research team plan to use an iterative approach (aka adaptive design); results and analysis from the first participants will be used to influence data collection moving forward for future participants (e.g. interview questions asked, timing and duration of biometric sensors being worn, etc.). See Section 4.0 for the definition of feasibility.

Note: The rationale for using telehealth is for human subjects' protections in the context of COVID-19 era infection control practices. Specifically, subject health care providers and study actors cannot currently meet inside in person without wearing masks. Masks will adversely affect the study of communication and emotion. Given that serious illness conversations are increasingly occurring by telehealth in the COVID-19 era, this scientific change could be considered a strength as the research team seeks to learn more about the exchangeability of telehealth for in-person clinical services.

Aim 2: Compare and test two wearable biometric sensors against wearable ECG chest band (gold standard) to evaluate reliability, accuracy, and ease of use from participant and investigator perspectives. The study purpose is to critically appraise the less expensive sensor versus the more expensive research model in different tasks (resting vs patient encounter vs interview) and over different domains (reliability, accuracy, ease of use). To compare the sensors, each participant will wear all three: (one on each arm and the chest band) during the encounter. The research team will define the benchmark for reliability as heart rate variability available ≥90% of the task against the gold standard (e.g. ECG chest band). The research team will use feedback from investigators and participants to grade ease of use. Accuracy will be measured in terms of the time-weighted absolute difference in resting heart rate variability between the consumer and the gold standard sensor.

Aim 3: Assess the correlation between study clinicians' documentation of serious illness conversations using an electronic template against independent expert review and documentation of the video-recorded and transcribed conversation.

Documenting serious illness conversations is an important way to record and share the patient's preferences, goals of care, and illness understanding with other clinicians. Embedded documentation tools, like a template, are common strategies to promote this documentation by reducing the labor to generate the documentation and encourages a uniform structure. Yet little is known about this process of translation - from what the patient says to what the clinician documents - specific to serious illness communication. By using a mixed-methods comparison of clinician-generated serious illness documentation to the transcribed conversations, the research team can perform an exploratory analysis of individual clinician and clinician specialty (e.g. palliative care, oncology) differences in the translation of the serious illness conversation into a documented note. Examples of correlation metrics that the research team may use include agreement and/or inter-rater reliability for closed-ended template items and narrative length and qualitative content analysis for open-ended template items between the study clinician and expert reviewer.

ELIGIBILITY:
Inclusion Criteria:

Clinicians who have been previously trained in the serious illness conversation guide. Two groups of participants will be recruited.

* hematology/oncology faculty
* specialty-trained palliative care clinicians

Exclusion Criteria:

* individuals who have a diagnosis of cardiovascular dysfunction

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Attending physicians in medical oncology or palliative care
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Investigator Assessed Feasibility of collecting clinician derived data on emotion regulation | Day 1
  This is a composite measure with four criteria: 1) >60% approached clinicians enroll on study; 2) <5% of missing time from encounter audio file; 3) <20% of missing time from heart rate variability collection; and 4) survey completion rates >90% of all items. All four criteria must be met for investigators to assess as feasible.

SECONDARY OUTCOMES:
The number of participants with heart rate variability data collected for more than 90% of the conversation task | Day 1
  time stamps for heart rate sensors and the HRV tracings used to determine time sensor collected HRV data
Completeness of Documentation | Day 1
  The documentation template clinicians are asked to use has 10 text fields they can complete. The study team will describe the number of fields each clinician completes. Qualitative analysis will assess content of text in those fields

CONTACTS AND LOCATIONS:
Overall Officials: Garrett T Wasp, MD, MPH, Principal Investigator — Dartmouth Cancer Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided